CLINICAL TRIAL: NCT02836769
Title: Development and Pilot Evaluation of Rehabilitation Consult for Survivors of Head and Neck Cancer
Brief Title: Development and Evaluation of Rehabilitation Consult for Survivors of Head and Neck Cancer
Acronym: HNC-RC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Princess Margaret Hospital, Canada (Other); Toronto General Hospital (Other); University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 246-2013
Record Dates: First submitted 2015-12-04; First posted 2016-07-19 (Estimated); Results first posted 2021-09-17 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-08

CONDITIONS: Head and Neck Neoplasms
Keywords: Rehabilitation; Head and neck cancer; Quality of life; self-efficacy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rehabilitation Consult (RC) (Experimental): Pilot testing: single group pre-post design
  Interventions: Behavioral: Rehabilitation Consult (RC)

INTERVENTIONS:
Behavioral: Rehabilitation Consult (RC) — The RC was designed to foster key contributors to self management in the participants. The RC is administered by a rehabilitation professional and consists of an initial one-hour face-to-face consult and follow-up appointment(s) 2-12 weeks later, either telephone or face-to-face. The initial consult consists of orientation, consultation, goal-setting, teaching cognitive strategies, introduction to online resources/action planning/planning coping responses, review/implementation intentions/scheduling follow-up. The follow-up consists of a reminder, reorientation, checking of progress on goals and plans, re-planning as necessary, and discharge or scheduling of further follow-up as necessary.

SUMMARY:
Although evidence exists to support cancer rehabilitation, services are fragmented and rehabilitation professionals are consulted infrequently and often long after treatment ends, when chronicity of problems limits the impact of intervention. Therefore, the objective of this project is to develop, implement, and conduct a pilot evaluation of the Rehabilitation Consult (RC). The RC program goals are to increase knowledge about rehabilitation needs and resources to meet those needs; to establish individualized rehabilitation goals for HNC survivors and personalized action plans to meet those goals; and to provide support to HNC survivors for the implementation and evaluation of action plans. This project consisted of intervention development and pilot evaluation; this trial registration describes the pilot evaluation phase only.

DETAILED DESCRIPTION:
A RC for survivors of head and neck cancer (HNC) was developed in collaboration with an Advisory Panel that includes survivors, family members, health care professionals, and health system representatives. This phase of the study aims to conduct a pilot evaluation of the RC using a mixed method, single group study with a convenience sample of approximately 35 survivors of HNC post primary cancer treatment, recruited from the Princess Margaret Cancer Center HNC clinics. In addition to the RC intervention, participants will be required to attend 3 research assessments (pre intervention, post intervention, and 1 month follow-up) that are a combination of face-to-face visits and telephone calls.

Quantitative data analysis will be exploratory and descriptive, and effect sizes will be calculated for all outcomes to help plan for a future, controlled trial. Means, standard deviations, and Cohen's d effect size will be calculated for normally distributed data. For non-normally distributed data, medians, ranges, and a nonparametric effect size r will be calculated. For qualitative analysis, all interviews will be audio recorded, transcribed verbatim, and analyzed using a two-phased, hybrid approach that is both deductive and inductive. Findings will be summarized and reported to the Advisory Panel, who will then make recommendations regarding any additional modifications to the RC. The research team will make final decisions about RC modifications and will finalize a version for future evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Adult survivors of HNC who have completed active treatment (surgery, radiation, chemotherapy or any combination thereof) within 1-18 months.

Exclusion Criteria:

* Lack of English fluency,
* Cognitive impairment, or concurrent major degenerative conditions likely to cause functional deterioration, and
* Known active cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-01; Primary Completion 2017-12 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara McEwen, PhD, Principal Investigator — Sunnybrook Research Institute, St. John's Rehab Program
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, Odette Cancer Centre, Toronto, Ontario
  - University Health Network, Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Study Protocol — http://www.implementationscience.com/content/10/1/6 — Publication of the initial project protocol
- Available data/document: Clinical Study Report — http://link.springer.com/article/10.1007%2Fs00520-015-3021-1 — Publication based on findings from focus groups used to create the intervention in this study

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rehabilitation Consult (RC)
Started | 35
Received Intervention | 30
Completed Post-test Assessment | 21
Completed | 20
Not Completed | 15
Not completed — Lost to Follow-up | 10
Not completed — Medical withdrawal | 2
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Rehabilitation Consult (RC)
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weeks post-treatment [Mean (Standard Deviation); unit: weeks] | 38.2 (22)
Had rehab goals [Count of Participants; unit: Participants] | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in Functional Assessment of Cancer Therapy - Head and Neck (FACT - H&N)
Description: Cancer-specific self-report measure of quality of life, higher scores indicate higher self-reported quality of life. Scores can range from 0 to 148. Changes in overall score as well as subsets will be evaluated for evidence of impact of intervention.
Time Frame: A) 1 week post-intervention, B) 1-2 months post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rehabilitation Consult (RC)
Number analyzed (Participants) | 30
score on a scale
  Mean difference (post - pre) | 3.1 (11.6)
  Mean difference (follow-up - pre) | 5.3 (12.3)

2. Primary Outcome: Change in Medical Outcome Short Form (36) Health Survey - (SF-36)
Description: Self-report quality of life questionnaire. Higher scores indicate a higher self-reported quality of life. The Physical Composite Score (PCS) and the Mental Composite Score (MCS) are reported. Scores range from 0 to 100 for each individual item on the scale. These scores are then converted into composite totals based on the scoring system provided with the outcome measure.
Time Frame: A) 1 week post-intervention, B) 1-2 months post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rehabilitation Consult (RC)
Number analyzed (Participants) | 30
score on a scale
  PCS - Mean difference (post - pre) | 3.5 (7.6)
  PCS - Mean Difference (follow-up - pre) | 6.7 (8.0)
  MCS - Mean difference (post - pre) | 4.3 (9.5)
  MCS - Mean Difference (follow-up - pre) | 2.8 (7.7)

3. Secondary Outcome: Change in Goal Performance, Satisfaction, and Self-efficacy
Description: Participants completed the Brief Rehabilitation Assessment for Survivors Of Head And Neck Cancer (BRASH), a self report tool where participants rate their current performance, satisfaction with self-selected rehab goals, and rate their confidence in their ability to achieve each goal. Higher scores indicate greater self-reported, performance, satisfaction, and self-efficacy. Scores for each of confidence, performance, and satisfaction can range from 0 to 100. Each category is then compared to itself and the change calculated by subtracting the earlier score from the latter.
Time Frame: A) 1 week post-intervention, B) 1-2 months post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rehabilitation Consult (RC)
Number analyzed (Participants) | 30
score on a scale
  Performance (post - pre) | 16.6 (32.3)
  Performance (follow-up - pre) | 37.3 (31.2)
  Satisfaction (post - pre) | 26.9 (35.4)
  Satisfaction (follow-up- pre) | 39.2 (32.6)
  Self-efficacy (post - pre) | 18.4 (27.1)
  Self-efficacy (follow-up- pre) | 17.1 (35.8)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the 15 months when study participants were enrolled.
Description: The risk of serious adverse events, mortality, and other adverse events was low because the study tested a behavioural intervention. Definitions of adverse events are in alignment with the Clinicaltrials.gov definitions.
Arm/Group | Rehabilitation Consult (RC)
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

LIMITATIONS AND CAVEATS:
This study did not include a control group and it is not known whether the improvements are due to the intervention, time, or other factors. Results from a single hospital may not be generalizable to other head and neck populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-11): https://cdn.clinicaltrials.gov/large-docs/69/NCT02836769/Prot_SAP_000.pdf